CLINICAL TRIAL: NCT03517306
Title: PET/CTbased Radiomics for Lung Cancer (PERL): a Retrospective Multi-center Study
Brief Title: PET/CT Based Radiomics for Lung Cancer (PERL)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Beijing Chao Yang Hospital (Other); General Hospital of Ningxia Medical University (Other); Soochow University (Other); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianhua Yan, Professor, Second Affiliated Hospital of Wenzhou Medical University
Other Study IDs: SAHoWMU-CR2018-05-223
Record Dates: First submitted 2018-04-19; First posted 2018-05-07 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Lung Cancer
Keywords: lung cancer, FDG, PET/CT, radiomics
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Beijing: No interventions
  Interventions: Other: No Interventions
- Ningxia: No interventions
  Interventions: Other: No Interventions
- Wenzhou: No interventions
  Interventions: Other: No Interventions
- Changzhou: No interventions
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No Interventions

SUMMARY:
The investigators investigate the utility of FDG PET/CT based radiomics in lung cancer, including diagnosis and prognosis.

DETAILED DESCRIPTION:
Recent studies have shown that, in addition to inter-tumor heterogeneity, tumors often display startling intratumoral heterogeneity in various features including histology, gene expression, genotype, and metastatic and proliferative potential, which is often associated with adverse tumor biology. Unfortunately, it is difficult to assess intratumoral heterogeneity with random sampling or biopsy as this does not represent the full extent of phenotypic or genetic variation within a tumor. Given the limitations of current biopsy strategies, there is an important potential for medical imaging, which has the ability to capture intratumoral heterogeneity in a non-invasive way.

Borrowed from the concept in genomics and/or proteomics, radiomics was specifically proposed for medical or radiological images. It is a promising technique for improving diagnosis, staging, prognosis, treatment response prediction and potentially allowing personalization of cancer treatment. It is a process of extraction and analysis of high-dimensional image features from radiological images obtained with CT, MR or PET, which could be either qualitative or quantitative. The basic assumption of radiomics is that tumor biology could be captured by radiomic features .

The purpose of this study is to investigate the utility of FDG PET/CT based radiomics in lung cancer. Four PET/CT centers will be involved in this study, in which more than 1000 patients diagnosed as lung cancer will be retrospectively enrolled.

ELIGIBILITY:
Inclusion Criteria:

- All patients diagnosed as lung cancer patients who had a FDG PET/CT scan before treatment between 1 Jan, 2013 and 30 December, 2016 in the four collaborative hospitals.

Exclusion Criteria:

- The patient without follow-up information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed as lung cancer patients who had a FDG PET/CT scan before treatment between 1 Jan, 2013 and 30 December, 2016 in the four collaborative hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-09-28 (Estimated)

PRIMARY OUTCOMES:
Creation of a FDG PET/CT based radiomic score for survival | Time Frame: 3 years
  Multiple quantitative radiomic features including SUV, metabolic volume, shape and texture will be measured from FDG PET/CT images. The all subjects will be randomly separated into a training and validation data. The multiple image features will be aggregated into a single combined radiomic score for survival with an appropriate machine learning method and the training data.

SECONDARY OUTCOMES:
Validation of a FDG PET/CT based radiomic score for survival | Time Frame: 3 years
  The created radiomic score developed in the primary outcome will be evaluated with the validation data in terms of survival(progress-free or overall survival)

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available to other researchers.